CLINICAL TRIAL: NCT00408239
Title: Factor Xa Inhibitor YM150 for Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement: A Randomized, Enoxaparin-controlled, Open Label, Dose-escalation Study
Brief Title: Factor Xa Inhibitor for Prevention of Venous Thromboembolism in Patients Undergoing Elective Total Knee Replacement
Acronym: PEARL-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 150-CL-029
Record Dates: First submitted 2006-12-04; First posted 2006-12-06 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Thromboembolism
Keywords: Factor Xa inhibitor; Thromboembolism; Arthroplasty; Knee Replacement; Prevention and Control
MeSH Terms: conditions — Thromboembolism | interventions — Enoxaparin

ARMS (3):
- 1 (Experimental): Dose regimen 1
  Interventions: Drug: YM150
- 2 (Active Comparator)
  Interventions: Drug: enoxaparin
- 3 (Experimental): Dose regimen 2
  Interventions: Drug: YM150

INTERVENTIONS:
Drug: YM150 — Oral
  Arms: 1; 3
Drug: enoxaparin — Sub cutaneous
  Arms: 2

SUMMARY:
Evaluate the safety and tolerability of escalating oral doses of YM150 in patients undergoing elective primary total knee replacement surgery

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for elective primary total knee replacement surgery
* Legal minimum age requirement ( country-specific)
* Written informed consent has been obtained

Exclusion Criteria:

* Documented history or considered to be at increased risk of venous thromboembolism
* Subjects considered to be at increased risk of bleeding:

  * Known hemorrhagic disorder and/or coagulation disorder
  * Thrombocytopenia
  * Clinically important bleeding occurred within 3 months prior to the screening visit
* Acute bacterial endocarditis
* Severe hypertension
* Retinopathy
* Concomitant use of anticoagulants / antiplatelet agents (including homeopathic drugs) and/or anticipated postoperative need for other reasons than prevention of DVT during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2006-12; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
All clinically relevant bleeds during treatment rated as major or clinically relevant non-major, and/or incidence of death due to any cause during study treatment | 2 Weeks

SECONDARY OUTCOMES:
Venous thromboembolism and/or bleeds | 2 Weeks
Other safety assessments | 2 Weeks
PK, PD variables | 2 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Chair — Astellas Pharma Inc
Locations (19):
- Jakarta, Indonesia
- Japan (7):
  - Chubu Region
  - Chugoku Region
  - Kansai Region
  - Kanto Region
  - Kyushyu Region
  - Shikoku Region
  - Tohoku Region
- Malaysia (2):
  - Kelantan
  - Kuala Lumpur
- Philippines (2):
  - Manila
  - Quezon City
- Singapore, Singapore
- South Korea (3):
  - Incheon
  - Jeonnam
  - Seoul
- Kaohsiung City, Taiwan
- Thailand (2):
  - Bangkok
  - Chiang Mai